CLINICAL TRIAL: NCT01731691
Title: Safety and Efficacy of Prolastin®-C (α1Proteinase Inhibitor, α1PI) in Human Immunodeficiency Virus-Infected Subjects
Brief Title: Safety and Efficacy of (α1Proteinase Inhibitor, α1PI) in HIV Disease
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Blinded review of the data suggested no significant diferences in outcomes.
Sponsor: Institute for Human Genetics and Biochemistry (Other)
Collaborators: AIDS Community Research Initiative of America (Other); Grifols Biologicals, LLC (Industry)
Responsible Party: Principal Investigator, Cynthia L Bristow, PhD, Principal Investigator, Institute for Human Genetics and Biochemistry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Prolastin-C in HIV disease
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Results first posted 2020-08-31 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: HIV Disease
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — alpha 1-Antitrypsin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- α1 Proteinase Inhibitor in HIV disease (Experimental): α1Proteinase Inhibitor (120mg/kg Prolastin-C) weekly for 8 weeks
  Interventions: Biological: α1 Proteinase Inhibitor
- Placebo in HIV disease (Placebo Comparator): Placebos weekly for 8 weeks
  Interventions: Drug: Placebos
- Uninfected controls (No Intervention): Blood collection only for 8 weeks

INTERVENTIONS:
Biological: α1 Proteinase Inhibitor — Prolastin-C treatment in HIV disease will be compared with placebo treatment in HIV disease and no treatment in uninfected volunteers.
  Other Names: Prolastin; Prolastin-C; Zemaira; Glassia
  Arms: α1 Proteinase Inhibitor in HIV disease
Drug: Placebos — Placebo treatment in HIV disease will be compared with Prolastin-C treatment in HIV disease and no treatment in uninfected volunteers.
  Other Names: Saline
  Arms: Placebo in HIV disease

SUMMARY:
Our primary objective is to further characterize the mechanism by which alpha-1PI regulates CD4 counts.

HIV-1 infected patients will be initiated on PROLASTIN®-C (Alpha-1 Proteinase Inhibitor [Human], Grifols Biotherapeutics Inc.) or placebo. Uninfected volunteers will be untreated and will be monitored for comparison.

DETAILED DESCRIPTION:
This study protocol is designed to investigate the benefit of a well-tolerated, FDA approved biological product that has been extensively used in a different patient population.

For more than 20 years, α1proteinase inhibitor (α1PI or α1antitrypsin) therapy has been the standard treatment for people with insufficient α1PI blood levels. This disorder, also known as α1antitrypsin deficiency, was previously thought to be caused only as an inherited trait due to the gene PIzz. Recent evidence shows that it can also be an acquired disease. Specifically, individuals with HIV-1 disease have been found to have severely low α1PI blood levels (Bristow et al., 2001; Bristow et al., 2010; Bristow et al., 2012). Many people with the inherited version of α1PI deficiency eventually develop emphysema, and among individuals with HIV-1 disease, 90% have acquired α1PI deficiency. Whether they go on to develop emphysema is still unresolved.

HIV-1 infected individuals are the first patient population identified so far in which severe α1PI deficiency is acquired through infection rather than being inherited.

It was found that a decrease in α1PI blood levels is directly correlated to a decrease in CD4 lymphocytes (Bristow et al., 2001; Bristow et al., 2012): In a pilot study to determine whether α1PI therapy might benefit the CD4 counts in HIV-1 infected patients (Clinicaltrials.gov NCT01370018), HIV-1 patients with infection-related α1PI deficiency received weekly α1PI therapy (120mg/kg) for a period of 8 weeks and results were compared with those of patients having the inherited version of α1PI deficiency who were simultaneously receiving weekly α1PI therapy (60mg/kg). None of the patients in the study had ever previously received α1PI therapy. It was found that CD4 cells rose to normal levels following 2 weeks of intravenous α1PI therapy with no adverse effects observed in the HIV-1 patients (n=3) or the control group of HIV-1 uninfected, α1PI deficiency patients (n=2). The new crop of CD4 cells were functional, capable of fighting infection, and appeared to be generated from bone marrow-derived stem cells (Bristow et al., 2010). As a bonus, it was found in the HIV-1 patients that LDL levels (bad cholesterol) decreased and HDL levels (good cholesterol) increased {Bristow et al., in review).

The information gained from the initial pilot study will be incorporated into this study design to further characterize the mechanism of lymphocyte renewal and to increase the number of patients observed. Only minor modifications to the pilot protocol are proposed including the sample size, addition of volunteers not receiving therapy, and a double-blind design: Ten (10) HIV-1 infected patients will be dosed with PROLASTIN®-C (Grifols Therapeutics Inc.), five (5) will be dosed with placebo, and five (5) uninfected volunteers not receiving therapy will be monitored.

It has been observed that CD4 counts and cholesterol levels are correlated and that there is cyclic variation in individuals with and without HIV. To examine whether there are differences due to HIV infection in cyclic variation of CD4 counts, cholesterol levels, and other values monitored during this study, five (5) volunteers, who do not have HIV, will be included in the study for blood collection only.

In a previous study, we determined that in individuals with abnormally low active α1PI levels, CD4 counts exhibit sinusoidal cycling with 23 day periodicity. Wave form appearance of CD4 cells with a peak every 23 days is a pattern that is indicative of adult thymopoiesis. We showed that in response to α1PI therapy, HIV infected and uninfected individuals exhibited an increased CD4 counts axis of oscillation, but no change in periodicity. In contrast, one uninfected individual who was not receiving therapy, exhibited no change in the axis of oscillation, but periodicity was 27 days. Human adult thymopoiesis is not well characterized, and based on these results, we have two hypotheses.

One hypothesis is that in response to α1PI therapy, thymopoiesis will increase, manifested by an increased axis of oscillation and increased numbers of recent thymic emigrants. In the proposed study, we will perform weekly TREC analysis which measures recent thymic emigrants and is definitive for thymopoiesis. We will test whether the changes in TREC numbers corresponds with changes in the CD4 counts axis of oscillation in HIV infected individuals receiving α1PI therapy as compared with HIV infected individuals with abnormally low active α1PI levels not on α1PI therapy, and HIV uninfected individuals with normal active α1PI levels not on α1PI therapy.

The second hypothesis is that in individuals with abnormally low active α1PI levels, the periodicity of CD4 counts is shorter than in individuals with normal active α1PI levels. Although we will measure periodicity in only 5 individuals with normal active α1PI levels and 15 with abnormal active α1PI levels, this will allow us to determine whether active α1PI is a linear determinate of periodicity or whether there are other variables that regulate periodicity. In an 8-week study, only 2 periods can be observed. Thus, following an 8-week regimen of therapy, one study subject may be asked to continue for a second 8-week regimen of therapy to allow the observation of 5 periods.

In addition to these two primary hypotheses regarding CD4 counts, we have found that HDL and LDL levels are linearly dependent on the balance of active and inactive α1PI levels (manuscript in review). This phenomenon is due the transport of HDL and LDL by CD4 cells. We found that in HIV infected individuals with abnormally low active α1PI and abnormally high inactive α1PI, HDL and LDL increased or decreased differently from individuals with normal active α1PI. Based on these results, our hypothesis is that in HIV infected individuals with abnormally low active α1PI receiving α1PI therapy, LDL levels will decrease and HDL levels will increase as active α1PI levels increase in contrast to HIV uninfected individuals with normal active α1PI levels not on therapy and in contrast to HIV infected individuals with abnormally low active α1PI levels not on therapy.

Prolastin-C treatment will be given weekly for eight (8) to sixteen (16) weeks by intravenous infusion. Blood will be collected immediately prior to each infusion. As in the previous study, complete blood count, lymphocyte phenotype, extended lymphocyte phenotype, lymphocyte function; HIV-1 viral load, lipid levels, blood chemistry, and markers of inflammation will be measured. The present study will also include measurements for HIV-1 tropism and markers for recent thymic emigrants.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 patients must have confirmed HIV-1 disease, diagnosed using the standard criteria and be on antiretroviral therapy. Uninfected volunteers will be age and gender matched.
2. HIV-1 patients must have measurable disease, defined as HIV-1 infected patients on antiretroviral therapy with undetectable HIV RNA (<1000 HIV RNA copies/ml) and CD4 counts more than 200 and less than 600 cells/uL.
3. Not have previously received α1PI augmentation therapy
4. Age at least 18 years and under 65 years
5. Capacity for and commitment to attend all protocol scheduled visits at ACRIA
6. Life expectancy of greater than 5 years
7. Patients must have lab values within the limits defined below:

   * WBC >4,1000/uL
   * ANC >1,000/uL
   * platelets >100,000//uL
   * total bilirubin 2-12 mg/dL
   * AST(SGOT)/ALT(SGPT) < or = 2.5 X upper limit of normal
   * creatinine Male : 0.50-1.30 mg/dL Female: 0.40-1.20 mg/dL
8. HIV-1 patients must have active α1PI below 11 uM (normal is 18-53 uM)
9. HIV-1 patients must have one year history (prior to the study) with CD4+ lymphocytes at levels greater than 200 and less than 400 cells/uL
10. HIV-1 patients must have absence of symptoms suggestive of HIV-1 disease progression
11. HIV-1 patients must have adequate suppression of virus (<400 HIV RNA/mL)
12. HIV-1 patients must have a history of compliance with antiretroviral medication based on undetectable virus levels
13. No evidence of malignancy
14. The effects of Prolastin-C on the developing human fetus at the recommended therapeutic dose are unknown: At any time throughout the study, from the signing of the informed consent form until after the last study visit, all female and male subjects who are biologically capable of having children must agree and commit to use a reliable method of birth control.
15. Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

1. Recent illness that will prevent the patient from participating in required study activities
2. Patients receiving other investigational agents
3. Patients with known malignancies
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Prolastin-C
5. IgA deficient patients
6. Patients with ≥1000 HIV-1 RNA copies/ mL
7. Patients with >600 CD4 cells/uL
8. Uncontrolled illness including, but not limited to, ongoing or active infection, myeloid dysplastic syndrome, anemia, bone marrow failure, DiGeorge Syndrome, thymic disorders, or psychiatric illness/social situations that would limit compliance with study requirements
9. Pregnant and breastfeeding women
10. Refusal to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bristow, PhD, Principal Investigator — Institute for Human Genetics and Biochemistry
Locations (1):
- ACRIA, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Incomplete data was made available to the PI.

REFERENCES:
- [Background] Bristow CL, Babayeva MA, LaBrunda M, Mullen MP, Winston R. alpha1Proteinase inhibitor regulates CD4+ lymphocyte levels and is rate limiting in HIV-1 disease. PLoS One. 2012;7(2):e31383. doi: 10.1371/journal.pone.0031383. Epub 2012 Feb 17. PMID 22363634
- [Background] Bristow CL, Patel H, Arnold RR. Self antigen prognostic for human immunodeficiency virus disease progression. Clin Diagn Lab Immunol. 2001 Sep;8(5):937-42. doi: 10.1128/CDLI.8.5.937-942.2001. PMID 11527807
- [Result] Bristow CL, Ferrando-Martinez S, Ruiz-Mateos E, Leal M, Winston R. Development of Immature CD4+CD8+T Cells Into Mature CD4+ T Cells Requires Alpha-1 Antitrypsin as Observed by Treatment in HIV-1 Infected and Uninfected Controls. Front Cell Dev Biol. 2019 Nov 21;7:278. doi: 10.3389/fcell.2019.00278. eCollection 2019. PMID 31824943

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Volunteers were recruited by ACRIA by placing advertisements in neighborhood publications. A total of 227 patients were interviewed as potential candidates. The first study candidate was screened on January 14, 2013 and the first HIV+ subject was randomized (treatment/placebo) on April 25, 2013.
Pre-assignment Details: Of the 21 potential subjects screened, 12 (57%) reached the baseline visit. All 12 were enrolled and all completed the study.
Period: Overall Study
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Started | 3 | 5 | 4
Completed | 3 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- α1 Proteinase Inhibitor in HIV Disease: α1Proteinase Inhibitor (120mg/kg Prolastin-C) weekly for 8 weeks
  α1 Proteinase Inhibitor: Prolastin-C treatment in HIV disease will be compared with placebo treatment in HIV disease and no treatment in uninfected volunteers.
  The subjects in the HIV+ groups (Prolastin-C and Placebo) were not comparable to those in the HIV- group.
- Placebo in HIV Disease: Placebos weekly for 8 weeks
  Placebos: Placebo treatment in HIV disease will be compared with Prolastin-C treatment in HIV disease and no treatment in uninfected volunteers.
  The subjects in the HIV+ groups (Prolastin-C and Placebo) were not comparable to those in the HIV- group.
- Uninfected Controls: Blood collection only for 8 weeks
  The subjects in the HIV+ groups (Prolastin-C and Placebo) were not comparable to those in the HIV- group.
- Total: Total of all reporting groups
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls | Total
Number analyzed (Participants) | 3 | 5 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 5 | 4 | 12
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (5) | 52 (7) | 32 (10) | 46 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 3
  Male | 2 | 4 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 4
  Not Hispanic or Latino | 3 | 3 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 5 | 4 | 12
CD4 [Mean (Standard Deviation); unit: cells/uL] | 365 (116) | 438 (108) | 651 (239) | 491 (193)
CD8 [Mean (Standard Deviation); unit: cells/uL] | 958 (340) | 872 (271) | 324 (53) | 711 (363)
CD4/CD8 Ratio [Mean (Standard Deviation); unit: Ratio] | 0.42 (0.17) | 0.53 (0.18) | 2.00 (0.58) | 0.99 (0.82)
α1 Proteinase Inhibitor [Mean (Standard Deviation); unit: uM] — Measured as active concentration, not as the traditional total concentration.
  uM | 14 (4) | 12 (6) | 21 (10) | 15 (8)
HDL [Mean (Standard Deviation); unit: mg/dL] | 55 (14) | 65 (14) | 58 (10) | 60 (12)
LDL [Mean (Standard Deviation); unit: mg/dL] | 89 (1.5) | 83 (16) | 83 (20) | 85 (14)

OUTCOME MEASURES:

1. Primary Outcome: CD4 Counts
Description: It has been observed that CD4 counts and cholesterol levels are correlated and that there is cyclic variation in individuals with and without HIV.
Time Frame: 9 weeks after initiation of treatment
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
cells/uL | 326 (103) | 437 (180) | 649 (141)

2. Primary Outcome: CD8
Description: as for outcome 1
Time Frame: 9 weeks after initiation of treatment
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
cells/uL | 848 (202) | 946 (365) | 302 (61)

3. Primary Outcome: CD4/CD8 Ratio
Description: as for outcome 1
Time Frame: 9 weeks after initiation of treatment
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
Ratio | 0.41 (0.18) | 0.48 (0.14) | 2.20 (0.55)

4. Primary Outcome: Alpha-1 Proteinase Inhibitor
Time Frame: weekly for 8 weeks
Measure: Mean (Standard Deviation); unit: micromol
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
micromol | 13.7 (3.4) | 13.6 (4.1) | 19 (9.5)

5. Primary Outcome: sj/betaTrec Ratio
Time Frame: weekly for 8 weeks
Measure: Mean (Standard Deviation); unit: sj/beta ratio
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
sj/beta ratio | 353.52 (353.54) | 271.19 (414.34) | 375.96 (357.81)

6. Primary Outcome: High Density Lipoprotein (HDL)
Time Frame: weekly for 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
mg/dL | 49.29 (6.21) | 63.14 (14.51) | 61.13 (10.40)

7. Primary Outcome: Low Density Lipoprotein (LDL)
Time Frame: weekly for 8 weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
Number analyzed (Participants) | 3 | 5 | 4
mg/dL | 90.67 (9.21) | 77.23 (25.19) | 75.19 (15.32)

ADVERSE EVENTS:
Time Frame: 9 weeks from initiation of therapy
Description: Zero patients experienced adverse events including in any of the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Zero adverse events resulted in life-threatening incidents or hospitalization or jeopardized the participant.
Arm/Group | α1 Proteinase Inhibitor in HIV Disease | Placebo in HIV Disease | Uninfected Controls
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/3 | 0/5 | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed; Technical problems with measurement leading to unreliable or uninterpretable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No